CLINICAL TRIAL: NCT05105685
Title: Effectiveness of Recombinant Human Growth Hormone Therapy for Children With Phelan-McDermid Syndrome: An Open-label, Cross-over, Preliminary Study
Brief Title: Effectiveness of Recombinant Human Growth Hormone Therapy for Children With PMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 395779225
Record Dates: First submitted 2021-10-25; First posted 2021-11-03 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Phelan-McDermid Syndrome; Growth Hormone Treatment
Keywords: Phelan-McDermid Syndrome; Growth Hormone Treatment; cross-over; Placebo-controlled
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome | interventions — Growth Hormone; Long-Term Synaptic Depression; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): Subjects were randomly divided into two different groups. Group A began with placebo while group B with rhGH. Randomisation of the treatment order (i.e., starting with rhGH or placebo) was done through a permuted four-block designed by the physician, who was the only one not blinded for treatment allocation.
  Interventions: Drug: Saline
- Group B (Experimental): Subjects were randomly divided into two different groups. Group A began with placebo while group B with rhGH. Randomisation of the treatment order (i.e., starting with rhGH or placebo) was done through a permuted four-block designed by the physician, who was the only one not blinded for treatment allocation.
  Interventions: Drug: recombinant human growth hormone

INTERVENTIONS:
Drug: recombinant human growth hormone — RhGH treatment was started at 0.1 IU/kg once daily
  Other Names: rhGH (Changchun Jinsai Pharmaceutical Co., Ltd, S20080011)
  Arms: Group B
Drug: Saline — Saline was started at 0.1 IU/kg once daily as the placebo
  Arms: Group A

SUMMARY:
In summary, this piot study with 6 participants shown that recombinant human growth hormone (rhGH) has a positive effect on the treatment with PMS. In addition, This study indicated that rhGH can improve PMS symptoms via increase the level of serum insulin-like growth factor-1 (IGF-1) and insulin-like growth factor binding protein 3 (IGFBP-3). RhGH may be low cost, more accessible, alternative treatment for PMS.

DETAILED DESCRIPTION:
Compared with the placebo, rhGH treatment significantly decreased the total scores and subscale scores of GDS (P <0.05), while the total scores and subscale scores of SC-ABC significantly decreased (P < 0.05) following three-months rhGH treatment. The similar results were also observed in comparison with baseline. Compared with the baseline, the level of serum IGF-1 and IGFBP-3 increased significantly (P < 0.05) following three-months rhGH treatment, while the placebo group had no significant impact on serum IGF-1 and IGFBP-3 (P > 0.05). One participant developed skin allergy the day after the first rhGH treatment, which were resolved later.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PMS aged from 1years to 5 years

Exclusion Criteria:

- active or suspected tumour, intracranial hypertension, chronic kidney disease, acute proliferative or severe nonproliferative diabetic retinopathy, allergy to rhGH or severe comorbidity

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
level of serum IGF-1 and IGFBP-3 | 3 months
  All laboratory indices were completed in the morning while the participants fasted and were analysed by the laboratory of the investigators' hospital.
Chinese version of the Gesell Development Scale (GDS) | 3 months
  To measure neuropsychological development. The development quotient (DQ) in the GDS was used to quantify neurodevelopment, which can indicate the level of neurodevelopment and is interpreted as follows: DQ=86 as normal, DQ 76 to 85 as marginally delayed, DQ at 55-75 as slightly delayed, DQ at 40 to 54 as moderately delayed, and DQ⩽39 as severely delayed.
Simplified Chinese version of the Aberrant Behavior Checklist (SC-ABC) | 3 months
  Different from its English version that created by Krug in 1980 , SC-ABC was based on the study of Krug in 2009, in which proved ABC can be used in 14 months children, then it was translated into Simplified Chinese by the researchers of Peking University Sixth Hospital. To date, the SC-ABC scale has been verified and widely used for more than 10 years to assess the changes of symptoms in Chinese children aged from 14 months to 14 years old with behavioral problems.
  This checklist includes 57 items and five subscales: sensory behavior, social relating, body and object use, language and communication skills, and social and adaptive skills. Each item was scored from 0 to 3,with higher scores indicate more severe symptoms.
Adverse events | 3 months
  Adverse events (AEs) were measured during the trial during via monitoring visits or phone calls using an adapted semi-structured interview every two weeks

CONTACTS AND LOCATIONS:
Overall Officials: YueYing Liu, Phd, Study Director — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of JiangNan University, Department of Pediatrics, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No